CLINICAL TRIAL: NCT05608343
Title: A Phase 3, Randomized, Double-Blind, Vehicle-Controlled, Multicenter Study to Assess the Efficacy and Safety of Difamilast Ointment 1% in Children, Adolescents, and Adults With Mild to Moderate Atopic Dermatitis
Brief Title: This Study is to Assess the Efficacy of Difamilast Ointment in Mild to Moderate Atopic Dermatitis(AD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Acrotech Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MM36-301
Record Dates: First submitted 2022-11-01; First posted 2022-11-08 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — difamilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Difamilast Ointment (Active Comparator): 1% Difamilast Ointment
  Interventions: Drug: Difamilast
- Vehicle Controlled (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Difamilast — Off-white ointment containing active ingredient, petrolatum and other ingredients
  Arms: Difamilast Ointment
Drug: Placebo — Matching Difamilast (Study drug) ointment without active ingradient
  Arms: Vehicle Controlled

SUMMARY:
This is a Phase 3 Double Blind multi-center study conducted at 40 investigational sites in United States to assess the efficacy and safety of Difamilast Ointment 1% in subjects ≥2 years of age with mild to moderate atopic dermatitis.

ELIGIBILITY:
Important Inclusion Criteria:

1. Subjects who are male or female ≥2 years of age
2. Subjects and/or their parent(s)/legal guardian(s) (if subject is under the legal age of consent) provide written informed consent in accordance with federal and/or local laws prior to the conduct of any study-related procedures.
3. Subjects who have a diagnosis of AD based on the American Academy of Dermatology AD diagnostic criteria
4. Subjects who have had a diagnosis of AD for at least 6 months prior to Screening visit
5. Subjects who have AD involvement ≥5% to ≤40% of treatable Body Surface Area (BSA) excluding scalp
6. Subjects who have an AD Severity of mild (2) or moderate (3) as measured by the IGA of AD Severity score at screening and baseline visit

Important Exclusion Criteria:

1. Female subjects who are pregnant or breastfeeding or who plan to become pregnant during the study and through 90 days after the last dose of study drug
2. Subjects who have evidence of spontaneous clearance of AD between screening and baseline visits
3. Subjects who have a history of unstable AD as assessed by the Investigator. Unstable AD is defined as disease flares occurring within 4 weeks prior to baseline visit
4. Subjects who have an active or acute skin infection (eg, herpes simplex, herpes zoster, and chicken pox) and/or clinically infected AD
5. Subject with greater than mild depression and suicidal ideation prior to screening or between screening and baseline visits
6. Subjects who have a known history of alcohol abuse or illicit drugs within 6 months prior to screening

Etc.,

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2023-10-27 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of twice-daily topical application of Difamilast ointment 1% compared to vehicle control in subjects ≥2 years of age with mild to moderate AD | Baseline, Day 29
  The proportion of subjects achieving success on the the 5-point Investigator Global Assessment (IGA) of AD Severity score at Day 29, and the success is defined as as a score of Clear (0) or Almost clear (1), with at least a 2-grade improvement from Baseline on the 5-point IGA of AD Severity score at Day 29

SECONDARY OUTCOMES:
To further characterize the efficacy of Difamilast ointment 1% compared to vehicle control in subjects with mild to moderate AD | Baseline, Day 15, Day 22 and Day 29
  The proportion of subjects achieving an IGA of AD Severity score of Clear (0) or Almost clear (1) at Day 29; the proportion of subjects achieving success on the 5-point IGA of AD Severity score at Day 22; the proportion of subjects achieving success on the 5-point IGA of AD Severity score at Day 15 The proportion of subjects achieving success on the 5-point IGA of AD Severity score at Day 22 The proportion of subjects achieving success on the 5-point IGA of AD Severity score at Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Uma Srinivas Atmuri, MPharm MS, Study Director — Acrotech Biopharma Inc.
Locations (39):
- United States (39):
  - AllerVie Health, Birmingham, Alabama
  - Elite Clinical Studies, LLC, Phoenix, Arizona
  - NEA Baptist Clinic-Dermatology, Jonesboro, Arkansas
  - First OC Dermatology, Fountain Valley, California
  - Center for Dermatology Clinical Research, Inc., Fremont, California
  - Antelope Valley Clinical Trials, Lancaster, California
  - Dermatology Research Associates, Los Angeles, California
  - Shahram Jacobs, MD Inc., Sherman Oaks, California
  - Clinical Trials Research Institute, Thousand Oaks, California
  - IMMUNOe Research Centers, Centennial, Colorado
  - TrueBlue Clinical Research, Brandon, Florida
  - Accel Research - Edgewater Clinical Research Unit, Edgewater, Florida
  - Tory Sullivan, MD PA, North Miami Beach, Florida
  - Nona Pediatrics, Orlando, Florida
  - Accel Research - Ormond Clinical Research Unit, Ormond Beach, Florida
  - Olympian Clinical Research, St. Petersburg, Florida
  - Arlington Dermatology, Rolling Meadows, Illinois
  - DS Research, Clarksville, Indiana
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - South Bend Clinic, South Bend, Indiana
  - DS Research, Louisville, Kentucky
  - Avant Research Associates, LLC, Crowley, Louisiana
  - Clinical Trials Management, LLC, Metairie, Louisiana
  - DermAssociates, LLC, Rockville, Maryland
  - Metro Boston Clinical Partners, Brighton, Massachusetts
  - Oakland Hills Dermatology, PC, Auburn Hills, Michigan
  - Minnesota Clinical Study Center, New Brighton, Minnesota
  - Dermatology Consulting Services, PLLC, High Point, North Carolina
  - Bexley Dermatology Research, Bexley, Ohio
  - Optima Research, Boardman, Ohio
  - Remington-Davis, Inc., Columbus, Ohio
  - Peak Research, LLC, Upper Saint Clair, Pennsylvania
  - International Clinical Research - Tennessee LLC, Murfreesboro, Tennessee
  - Arlington Research Center, Inc., Arlington, Texas
  - North Texas Center for Clinical Research, Frisco, Texas
  - Center for Clinical Studies, Ltd, LLP, Houston, Texas
  - Houston Center for Clinical Research, Sugar Land, Texas
  - Premier Clinical Research, LLC, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No